CLINICAL TRIAL: NCT05658393
Title: The Effect of a Mobile Health Application Developed for Patients With Liver Cirrhosis on Patient Activation, Self-Efficacy, and Quality of Life
Brief Title: Web-based Mobile Health Application for Patients With Liver Cirrhosis (ReLiver-N App)
Acronym: ReLiver-NApp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ferya Celik, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Akdeniz U
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Mobile Health; Liver Cirrhosis; Patient Activation
Keywords: liver cirrhosis; mobile health; Patient Activation
MeSH Terms: conditions — Liver Cirrhosis; Patient Participation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be divided into groups according to the randomization list created to assign each patient to a group. Two independent researchers will conduct the assignment of participants to the ReLiver-N App and active control groups and the evaluation of outcome measurement data. Researchers will not be blinded as they make these interventions. However, participants will be blinded because they do not know which group, they are in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ReLiver-N App Group (Experimental): The ReLiver-N App will be introduced to the participants with liver cirrhosis during face-to-face interviews. The ReLiver-N App group will have access to all the contents of the ReLiver-N App, which includes the "about us", "patient education information about liver cirrhosis ", "patient activity skills", and "measuring tools". During the follow-up period, the participants in the ReLiver-N App group will take WhatsApp messages once a week and be reminded to use the education program. The ReLiver-N App will be asked to use it for three months on daily and weekly inputs their results. During the follow-up period, the participants can contact researcher via the 24/7 on the ReLiver-N App. The clinical researchers of the team will answer the participant' questions via WhatsApp. Participants in the ReLiver-N group will also receive routine patient education and routine hospital follow-ups given by the Gastroenterology team.
  Interventions: Behavioral: ReLiver-N App
- Active Control Group (Active Comparator): The ReLiver-N App will be introduced to the participants with liver cirrhosis in the active control group during face-to-face interviews. The active control group will have access to only these fields "about us", "patient activity skills", and "measuring tools". Participants in the active control group will also receive routine patient education and routine hospital follow-ups given by the Gastroenterology team during the three-month follow-up period.
  Interventions: Behavioral: ReLiver-N App

INTERVENTIONS:
Behavioral: ReLiver-N App — Web-based mobile health application for patients with liver cirrhosis

SUMMARY:
This study evaluates the effect of a web-based mobile health application for patients with liver cirrhosis (ReLiver-N App) developed for enhancing patients' activation on the level of patient activation, self-efficacy, and quality of life. To manage liver cirrhosis after discharge, patients must continue to do some interventions at home like weight measurement, edema evaluation, and taking medications. To achieve this, the patient's activation level should be enhanced and that can contribute to hepatic rehabilitation. It would be beneficial to develop a web-based mobile health application for patients with liver cirrhosis that can enhance patient activation levels. The investigators developed the ReLiver-N App based ADDIE which is instructional design framework and created its contents of it. Our content includes about us, patient education information about liver cirrhosis, patient activity skills and measuring tools. Ten experts evaluated the quality of the content and the investigators conducted a feasibility test with three patients to assess the usability of the ReLiver-N App. A single-blind randomized controlled trial design will be applied. Patients with liver cirrhosis will be pretested and randomized (intervention (ReLiver-N App): 26, active control: 26) to the ReLiver-N App group and active control group. Both the ReLiver-N App group and active control group will use the ReLiver-N App for three months. While participants in the ReLiver-N group can reach all content of the ReLiver-N App. Participants in the active control group will have access to "about us", "patient activity skills", and "measuring tools" in the ReLiver-N App. Patient education information about liver cirrhosis will be encrypted.

DETAILED DESCRIPTION:
Liver cirrhosis is an important health problem that leads to morbidity and mortality. To maintain symptom management after discharge, patient education and activation should be enhanced. The unmet educational needs of patients with liver cirrhosis cause ineffective management of liver cirrhosis. It is important for patients to actively participate in patient activation practices and develop their skills. Patient activation practices, which are the responsibility of the patient in the management of liver cirrhosis, are easy to apply and provide effective results. Improving patient activation could help with early symptom detection and control of symptoms, and that can contribute to hepatic rehabilitation. It seems that using accessible and sustainable mobile health applications could help provide patient education and enhance activation. Mobile health applications make it possible to enable patients to provide information to enhance their level of activation. Mobile health applications developed for patient activation could help patients learn their responsibilities for health and be motivated to do them. When the level of patient activation gets higher, patients' self-efficacy and quality of life getting higher. The study evaluates the effect of the web-based mobile health application (ReLiver-N App) developed for patient activation in patients with liver cirrhosis on patient activation, self-efficacy, and quality of life.

Objective: It is aimed to develop a web-based mobile health application (ReLiver-N App) for patients with liver cirrhosis and to evaluate the effect of ReLiver-N App use on patients' activation, self-efficacy, and quality of life. The ReLiver-N App engages and supports patients with liver cirrhosis by increasing patient activation through m-health education. This could increase patient activation, self-efficacy, and quality of life. This study primarily aims the analysis the efficacy of ReLiver-N App on increasing patient activation, self-efficacy, and quality of life.

Method: The first stage of this study was the development stage of the ReLiver-N App based ADDIE which is instructional design framework. This stage included reading the content and designing the ReLiver-N App. The content of the ReLiver-N App was based on the needs of patients, evidence, and recommendations for patient education in liver cirrhosis such as guidelines, meta-analyses, randomized controlled trials, reliable patient education websites, and expert opinions. The investigators created the contents of the ReLiver-N App. Our content includes "about us", "patient education information about liver cirrhosis ", "patient activity skills", and "measuring tools". Patient education information topics include a healthy lifestyle, let's learn about liver cirrhosis, complications of liver cirrhosis, diagnosis, treatment methods, and let's enhance quality of life and self-efficacy. Patient activity skills are divided into two groups: daily activity skills and weekly activity skills. Daily activity skills include weight measurement, edema evaluation, and taking medications. Weekly activity skills include taking blood pressure, heart rate, and body temperature. Measurements questionnaires include pre-test, follow-up and end-point questionnaires. The participants can answer these questionnaire via ReLiver-N App. After preparing the content, 10 experts evaluated the quality of the content and the investigators conducted a feasibility test with three patients to assess the usability of the ReLiver-N App group.

In the second stage, the investigators will conduct a single-blind randomized controlled study to determine the effect of the ReLiver-N App developed for patients with liver cirrhosis on patient activation, self-efficacy, and quality of life. This study will be conducted in patients with liver cirrhosis who are followed up and treated in the Gastroenterology Outpatient Clinic and Inpatient Clinic and meets the inclusion criteria of the sample. In this study, the sample size was calculated based on 80% power and a 5% confidence interval on the G*POWER software package. The study will be conducted in patients with liver cirrhosis (n=52), 26 in the ReLiver-N App group and 26 in the control group. The patients who had been diagnosed with liver cirrhosis, were over 18 years of age, literate, had Child-Pugh Score A and B, had internet at home and a smartphone, consented to participate in the study and had no other psychiatric or emotional problems, language or cognitive difficulties, and barriers to verbal or written communication were included. It will be prepared in line with the Consolidated Standard of Reporting Trials - CONSORT 2018 guidelines. There will be a screening, pre-test at baseline, randomization, and follow-up.

Full sociodemographic, and clinical assessments and obtained consent will be carried out at the screening. At the screening stage, all participants will be informed about ReLiver-N App and this study face-to-face at the hospital first. After that participants could be used ReLiver-N App at home. The pre-test will be carried out baseline measurement. After baseline measurements will be undertaken by the researcher before randomization takes place.

A single-blinded randomized controlled trial is planned. An independent researcher who was not involved in the research will be assigned to the ReLiver-N App and active control groups with the web-based randomization program. Randomization will be done in https://www.randomizer.org/. Participants will be randomized 1:1 to the ReLiver-N App group and active control group. The ReLiver-N App group will have access to all the content of the ReLiver-N App, which includes the "about us", "patient education information about liver cirrhosis ", "patient activity skills", and "measuring tools". Passwords will be defined so that patients in the ReLiver-N App group can access the "patient education information about liver cirrhosis ". ReLiver-N App will be delivered face-to-face at the hospital first by the researcher, after that participants could be used it at home. Participants in the active control group will only have access to the "about us", "patient activity skills " and the "measuring tools" in the ReLiver-N App. Other fields will be encrypted. Patients in the active control group will also be informed about the area they can access. The ReLiver-N App will be asked to use it for three months on daily and weekly input their results like weight measurement, edema evaluation, and taking medications. The investigators will send a message to participants in the ReLiver-N group in a every week via Whatsapp to remind their patient activity skills. The participants were blinded because they were unaware of their randomization status. Since the researchers conducted the interventions, it is not possible to blind the researcher cause of the nature of the study.

Our primary outcomes are patient activation, self-efficacy, and quality of life. Outcomes will be measured at baseline and follow-up occurring 1, 2, and 3, months after enrolment. The hypotheses are as below:

It is hypothesized that compared with those receiving standard care after controlling for baseline levels, participants receiving the ReLiver-N App intervention will report significantly.

1. Participants receiving the ReLiver-N App intervention will have higher levels of patient activation than those receiving standard care after controlling for baseline levels of patient activation.
2. Participants receiving the ReLiver-N App intervention will have higher levels of self-efficacy than those receiving standard care after controlling for baseline levels of self-efficacy.
3. Participants receiving the ReLiver-N App intervention will have higher levels of quality of life than those receiving standard care after controlling for baseline levels of quality of life.

The investigators will evaluate outcomes by using the Patient Activation Measure (PAM), Self-Efficacy for Managing Chronic Disease 6-Item Scale, and Chronic Liver Disease Questionnaire (CLDQ).

Primary Outcome Measures Patient Activation Measure (PAM) The Patient Activation Measure (PAM) gauges a patient's level of belief, knowledge, skill, and self-assurance. 13 components make up the Patient Activation Measure. Patients are actively/successfully managing their disease when they receive higher scores on the scale. Each response option has a 4-point Likert scale with the options ranging from totally disagree to totally agree and 'non-applicable.' Scores for activities range from 0 to 100. Level 1, the lowest activity with a score of 47, deals with the idea that playing an active part is important. Level 2, which ranges from 47 to 55, denotes knowledge and the capacity for action. Level 3, which ranges from 55 to 72, deals with action. The highest activity, Level 4, with scores of >72.5, is keeping to a schedule even when under stress. Cronbach's alpha value of the original scale was determined as 0.88.

Self-Efficacy for Managing Chronic Disease 6-Item Scale The scale is scored on a scale of 1 to 10, with 1 being "not at all confident" and 10 being "totally confident." High scores on the scale denote high self-efficacy. The scale's score is the average of the six components. The lower score is taken into account in the computation if there are several responses to a question and the items are consecutive. This item is not included in the calculation if the two answers provided are not sequential. There must be at least 4 responses for the scale to be calculated. Cronbach's alpha value of the original scale was determined as 0.88.

Chronic Liver Disease Questionnaire The Chronic Liver Disease Questionnaire is a 29-item self-report questionnaire, consisting of six subdimension, which include abdominal symptoms, fatigue, systemic symptoms, activity, emotional function, and anxiety. All items ask for the symptoms during the previous two weeks. The overall ICC value of the original CLDQ is 0.59.

Conclusion: The ReLiver-N App is based on getting increase patient activation. It is expected that the ReLiver-N App will improve patient activation, self-efficacy, and quality of life. This study could contribute to the innovation of health care through the development of a new digital tool for patient education and activation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with liver cirrhosis
* Had Child-Pugh A and B categories
* 18 years of age or older
* No barriers to verbal or written communication
* Having internet at home and a smartphone Patients who consented to participate in the study.

Exclusion Criteria:

* Had Child-Pugh C category
* Had pregnant
* Liver transplanted
* Diagnosed with hepatocellular carcinoma
* Having dementia
* Having been diagnosed with a psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-07-09 (Actual)

PRIMARY OUTCOMES:
Patient Activation Measure (PAM) | Change from baseline PAM at one month, Change from baseline PAM at two months, Change from baseline PAM at three months
  The Patient Activation Measure (PAM) gauges a patient's level of belief, knowledge, skill, and self-assurance. 13 components make up the Patient Activation Measure. Patients are actively/successfully managing their disease when they receive higher scores on the scale. Each response option has a 4-point Likert scale with the options ranging from totally disagree to totally agree and 'non-applicable.' Scores for activities range from 0 to 100. Level 1, the lowest activity with a score of 47, deals with the idea that playing an active part is important. Level 2, which ranges from 47 to 55, denotes knowledge and the capacity for action. Level 3, which ranges from 55 to 72, deals with action. The highest activity, Level 4, with scores of >72.5, is keeping to a schedule even when under stress. Cronbach's alpha value of the original scale was determined as 0.88.
Self-Efficacy for Managing Chronic Disease 6-Item Scale (SEMCD6IS) | Change from baseline SEMCD6IS at one month, Change from baseline SEMCD6IS at two months, Change from baseline SEMCD6IS at three months
  The scale is scored on a scale of 1 to 10, with 1 being "not at all confident" and 10 being "totally confident." High scores on the scale denote high self-efficacy. The scale's score is the average of the six components. The lower score is taken into account in the computation if there are several responses to a question and the items are consecutive. This item is not included in the calculation if the two answers provided are not sequential. There must be at least 4 responses for the scale to be calculated. Cronbach's alpha value of the original scale was determined as 0.88.
Chronic Liver Disease Questionnaire (CLDQ) | Change from baseline CLDQ at one month, Change from baseline CLDQ at two months, Change from baseline CLDQ at three months
  The Chronic Liver Disease Questionnaire (CLDQ) is a 29-item self-report questionnaire, consisting of six subdimension, which include abdominal symptoms, fatigue, systemic symptoms, activity, emotional function, and anxiety. All items ask for the symptoms during the previous two weeks. The overall ICC value of the original CLDQ is 0.59.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It can be shared privately if other researchers would like to get it.